CLINICAL TRIAL: NCT05077332
Title: Leidos-Enabled Adaptive Protocol for Clinical Trials (LEAP-CT) to Evaluate the Safety and Efficacy of Drug Combinations in COVID-19 Patients
Brief Title: LEAP-CT for Treatment of COVID-19 Patients (Master Protocol)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Leidos Life Sciences (Industry)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LDOS-21-001
Record Dates: First submitted 2021-10-07; First posted 2021-10-14 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-12

CONDITIONS: 2019 Novel Coronavirus Disease; 2019 Novel Coronavirus Infection; 2019-nCoV Disease; 2019-nCoV Infection; COVID-19 Pandemic; COVID-19 Virus Disease; COVID-19 Virus Infection; Covid19; Coronavirus Disease 2019; SARS-CoV-2 Infection; SARS-CoV-2 Acute Respiratory Disease; COVID-19
Keywords: COVID-19; COVID; COVID19; SARS-CoV-2
MeSH Terms: conditions — COVID-19 | interventions — Famotidine; Celecoxib

STUDY DESIGN:
Intervention Model Description: Subjects randomized 1:1, study drug:placebo
Who Masked: Participant, Care Provider, Investigator
Masking Description: Only the participant is blinded in LDOS-21-001-01 (Addendum #1; inpatient study); All are blinded in LDOS-21-001-02 (Addendum #2; outpatient study).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Study Product) (Experimental): Participants will receive 80 mg famotidine (PO) QID and 400 mg celecoxib as a first dose, followed by 200 mg (PO) BID celecoxib, for 5 days. Following this 5-day period, participants will continue their famotidine treatment for an additional 9 days.
  Interventions: Drug: Famotidine; Drug: Celecoxib
- Group 2 (Reference Therapy) (Placebo Comparator): Participants will receive matching placebos QID and BID, for 5 days. Following this 5-day period, subjects will continue to receive matching famotidine placebo, QID, for an additional 9 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Famotidine — 80 mg tablet, QID for 14 days
  Other Names: Pepcid
  Arms: Group 1 (Study Product)
Drug: Celecoxib — 400 mg (initial dose) then 200 mg capsule, BID for 5 days
  Other Names: Celebrex
  Arms: Group 1 (Study Product)
Other: Placebo — tablet, QID for 14 days; capsule, BID for 5 days
  Arms: Group 2 (Reference Therapy)

SUMMARY:
This master protocol serves as a common reference for the inpatient and outpatient clinical studies that share common elements.

DETAILED DESCRIPTION:
There are currently two addenda to this master protocol:

Addendum 1, Study LDOS-21-001-01, is a Phase 2, randomized, single-blind, placebo-controlled study to evaluate the safety and efficacy of the combination of famotidine and celecoxib as a treatment in moderate-to-severe patients hospitalized for COVID-19.

Addendum 2, Study LDOS-21-001-02, is a Phase 2 randomized, placebo-controlled, double-blind study to evaluate the safety and efficacy of the combination of famotidine and celecoxib as a post-exposure prophylaxis (PEP) for newly infected COVID-19 patients.

ELIGIBILITY:
* For eligibility criteria specific to the protocol, see:
* Addendum #1 (LDOS-21-001-01) or
* Addendum #2 (LDOS-21-001-02)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2021-12-29 (Actual); Primary Completion 2025-11-10 (Actual); Study Completion 2025-11-10 (Actual)

PRIMARY OUTCOMES:
(LDOS-21-001-01) Time-to-event to achieve WHO level ≤3 | 30 days
  Evaluation of the time-to-event to achieve a WHO level score ≤3
(LDOS-21-001-01) All-Cause Mortality rate | 30 days
  Measured in whole numbers by participants removed from the study with reason of "death" in the electronic data capture system
(LDOS-21-001-02) Number of patients with at least one COVID-19-related medically attended contact due to increased COVID-19 symptom severity | 30 days
  Medically attended contact will be measured in whole numbers and reported as "1 medically attended contact" each time, in the electronic data capture system for all study participants
(LDOS-21-001-02) Number of patients with at least one COVID-19-related medically attended contact due to death (all-cause mortality) | 30 days
  Medically attended contact will be measured in whole numbers and reported as "1 medically attended contact" in the electronic data capture system for all study participants.

CONTACTS AND LOCATIONS:
Overall Officials: Brian A Roberts, MS, PMP, Study Director — Leidos, Inc.
Locations (1):
- US02-04: Integrated Health Solutions, Miami, Florida, United States

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Background] Malone RW, Tisdall P, Fremont-Smith P, Liu Y, Huang XP, White KM, Miorin L, Moreno E, Alon A, Delaforge E, Hennecker CD, Wang G, Pottel J, Blair RV, Roy CJ, Smith N, Hall JM, Tomera KM, Shapiro G, Mittermaier A, Kruse AC, Garcia-Sastre A, Roth BL, Glasspool-Malone J, Ricke DO. COVID-19: Famotidine, Histamine, Mast Cells, and Mechanisms. Front Pharmacol. 2021 Mar 23;12:633680. doi: 10.3389/fphar.2021.633680. eCollection 2021. PMID 33833683
- [Background] Janowitz T, Gablenz E, Pattinson D, Wang TC, Conigliaro J, Tracey K, Tuveson D. Famotidine use and quantitative symptom tracking for COVID-19 in non-hospitalised patients: a case series. Gut. 2020 Sep;69(9):1592-1597. doi: 10.1136/gutjnl-2020-321852. Epub 2020 Jun 4. PMID 32499303
- [Background] Hogan Ii RB, Hogan Iii RB, Cannon T, Rappai M, Studdard J, Paul D, Dooley TP. Dual-histamine receptor blockade with cetirizine - famotidine reduces pulmonary symptoms in COVID-19 patients. Pulm Pharmacol Ther. 2020 Aug;63:101942. doi: 10.1016/j.pupt.2020.101942. Epub 2020 Aug 29. PMID 32871242
- [Background] Tomera K, Malone R, Kittah J. Hospitalized COVID-19 Patients Treated with Celecoxib and High Dose Famotidine Adjuvant Therapy Sow Significant Clinical Responses. Frontiers in Pharmacology. 2021.
- [Background] Sun C, Chen Y, Hu L, Wu Y, Liang M, Ayaz Ahmed M, Bhan C, Guo Z, Yang H, Zuo Y, Yan Y, Zhou Q. Does Famotidine Reduce the Risk of Progression to Severe Disease, Death, and Intubation for COVID-19 Patients? A Systemic Review and Meta-Analysis. Dig Dis Sci. 2021 Nov;66(11):3929-3937. doi: 10.1007/s10620-021-06872-z. Epub 2021 Feb 24. PMID 33625613
- [Background] Shoaibi A, Fortin SP, Weinstein R, Berlin JA, Ryan P. Comparative Effectiveness of Famotidine in Hospitalized COVID-19 Patients. Am J Gastroenterol. 2021 Apr;116(4):692-699. doi: 10.14309/ajg.0000000000001153. PMID 33982938
- [Background] Sander WJ, O'Neill HG, Pohl CH. Prostaglandin E2 As a Modulator of Viral Infections. Front Physiol. 2017 Feb 14;8:89. doi: 10.3389/fphys.2017.00089. eCollection 2017. PMID 28261111
- [Background] Morimoto K, Shirata N, Taketomi Y, Tsuchiya S, Segi-Nishida E, Inazumi T, Kabashima K, Tanaka S, Murakami M, Narumiya S, Sugimoto Y. Prostaglandin E2-EP3 signaling induces inflammatory swelling by mast cell activation. J Immunol. 2014 Feb 1;192(3):1130-7. doi: 10.4049/jimmunol.1300290. Epub 2013 Dec 16. PMID 24342806
- [Background] Hong W, Chen Y, You K, Tan S, Wu F, Tao J, Chen X, Zhang J, Xiong Y, Yuan F, Yang Z, Chen T, Chen X, Peng P, Tai Q, Wang J, Zhang F, Li YX. Celebrex Adjuvant Therapy on Coronavirus Disease 2019: An Experimental Study. Front Pharmacol. 2020 Nov 6;11:561674. doi: 10.3389/fphar.2020.561674. eCollection 2020. PMID 33312125
- [Background] Chen JS, Alfajaro MM, Chow RD, Wei J, Filler RB, Eisenbarth SC, Wilen CB. Non-steroidal anti-inflammatory drugs dampen the cytokine and antibody response to SARS-CoV-2 infection. J Virol. 2021 Mar 10;95(7):e00014-21. doi: 10.1128/JVI.00014-21. Epub 2021 Jan 13. PMID 33441348